CLINICAL TRIAL: NCT04952454
Title: Non-endoscopic Endonasal, Transcanalicular, or External Dacryocystorhinostomy for Functional Epiphora: Which is Better?
Brief Title: Functional Epiphora Management Via Different Dacryocystorhinostomy (DCR) Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Can Ozturker, Asist. Prof., Istanbul University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1533-2020
Record Dates: First submitted 2021-07-01; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Functional Epiphora (Tearing Without Any Anatomical Block)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- External DCR (Active Comparator): Patients treated with External DCR for functional epiphora
  Interventions: Procedure: External Dacryocystorhinostomy
- Endonasal DCR (Active Comparator): Patients treated with Endonasal DCR for functional epiphora
  Interventions: Procedure: Endonasal Dacryocystorhinostomy
- Transcanalicular DCR (Active Comparator): Patients treated with Transcanalicular DCR for functional epiphora
  Interventions: Procedure: Transcanalicular Dacryocystorhinostomy

INTERVENTIONS:
Procedure: External Dacryocystorhinostomy — The resistance of the lacrimal drainage is lowered by creating a new ostium between the lacrimal sac and nasal cavity via skin incision.
  Arms: External DCR
Procedure: Endonasal Dacryocystorhinostomy — The resistance of the lacrimal drainage is lowered by creating a new ostium between the lacrimal sac and nasal cavity via endonasal route.
  Arms: Endonasal DCR
Procedure: Transcanalicular Dacryocystorhinostomy — The resistance of the lacrimal drainage is lowered by creating a new ostium between the lacrimal sac and nasal cavity via transcanalicular route.
  Arms: Transcanalicular DCR

SUMMARY:
135 eyes of 135 patients treated between 2005 and 2017 will be included in this study. The diagnosis of functional epiphora was made based on a patent lacrimal system with a delay in the fluorescein dye disappearance test (FDDT) or dacryoscintigraphy (DSG) without any ocular surface or eyelid abnormalities. The absence of epiphora and normalization of FDDT postoperatively was defined as success. The study's hypothesis is that external DCR with a suitable technique will have better results compared to endonasal and transcanalicular DCR

ELIGIBILITY:
Inclusion Criteria:

* patent lacrimal irrigation and delay in the lacrimal transit time demonstrated by fluorescein dye disappearance test (FDDT) or a dacryoscintigraphy (DSG)

Exclusion Criteria:

* Dry eye (tear break up time less than 10 seconds), ocular surface disorders, eyelid malposition or laxity, orbicularis weakness, partial block or stenosis of the lacrimal drainage, history of previous nasal, lacrimal, or ophthalmic surgeries, and a postoperative follow-up time less than six months

Min Age: 21 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who report resolution of theri tearing and normalization of fluorescein dye disappearance test. | Last follow-up time, approximately 6 months

SECONDARY OUTCOMES:
Number of patients who have continuing epiphora after the surgery with an anatomically blocked tear duct. | Last follow-up time, approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Can Ozturker, MD, Study Director — Istanbul University, Istanbul Facukty Of Medicine
Locations (2):
- McMaster University, Hamilton, Ontario, Canada
- Beyoglu Eye Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No